CLINICAL TRIAL: NCT07235436
Title: Cryopreservation of Platelets for Prophylactic Use in Onco-haematology: an in Vitro Study
Brief Title: Platelet Cryopreservation
Acronym: PLT-CRIO
Status: Completed | Type: Observational
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Other Study IDs: 1221/2020/TESS/IRCCSRE
Record Dates: First submitted 2025-09-17; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-09

CONDITIONS: Platelet Cryopreservation
Keywords: onco-hematological patient; cryopreservation; transfusion; platelets

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

SUMMARY:
The study "Cryopreservation of Platelets for Prophylactic Use in Onco-Hematology: an in vitro Study", coordinated by Dr. Lucia Merolle at the Department of Transfusion Medicine of the Azienda USL-IRCCS of Reggio Emilia, aims to investigate the impact of cryopreservation methods on platelet functionality and metabolism. The primary objective of this project is to determine the effects of cryogenic storage on platelet function. The study design involves the recruitment of donors, preparation of platelet concentrates, and their cryopreservation. After thawing, the products undergo a series of biochemical and functional evaluations, including platelet count, pH measurement, pro-inflammatory cytokine levels, morphological assessment, and activity testing. Data will then be analyzed to determine the minimal effective concentration required for safe and effective use. Platelet apheresis samples are collected and analyzed. Participation is proposed to platelet donors at the Department of Transfusion Medicine, and inclusion requires the signing of written informed consent, while refusal to provide consent will exclude individuals from the study.

DETAILED DESCRIPTION:
Platelets are essential blood components with pivotal roles in both hemostasis and inflammation. Thrombocytopenia, defined as a reduction in circulating platelet count, may result from impaired bone marrow production, increased consumption, splenic sequestration, or bleeding episodes, and is commonly managed through platelet transfusions aimed at restoring adequate counts and, when necessary, controlling hemorrhage. In clinical practice, the majority of platelet transfusions are administered to thrombocytopenic cancer patients with a prophylactic intent, where the primary requirement is sustained platelet survival to minimize the number of transfusions. Conversely, in actively bleeding patients, platelet transfusions are expected to provide rapid and efficient hemostasis, while their circulation time is of lesser relevance. Currently, platelet concentrates are stored at room temperature (22-24 °C) under continuous agitation for up to five days, after which they are discarded if unused. This storage method carries the risk of bacterial contamination and induces metabolic and structural changes that compromise platelet function, a phenomenon known as platelet storage lesion (PSL). Furthermore, the short shelf life limits the availability of platelets in emergency settings, as observed during the SARS-CoV-2 pandemic, when the demand for prophylactic platelet transfusions remained constant while supply was severely strained. In response, the Transfusion Medicine Unit in Reggio Emilia introduced cryopreservation of platelet concentrates to prevent future shortages. Cryopreservation allows storage of platelets for up to two years, offering an attractive alternative to conventional methods, not only extending storage duration but also reducing the risl of bacterial contamination. Although recent studies have demonstrated the safety and efficacy of cryopreserved platelets in bleeding patients, limited evidence exists for their use in prophylaxis among onco-hematologic patients. Major concerns include the potential for exacerbating thrombotic risk in patients with chronic hypercoagulability and the release of bioactive molecules such as growth factors and pro-inflammatory cytokines during thawing, which could have pro-tumorigenic effects. Platelet-tumor interactions are known to be complex, exerting both pro- and anti-tumoral influences, with the balance often favoring tumor progression. The present study therefore aims to evaluate the impact of cryopreservation on platelet functionality, structure and morphology, as well as to assess potential pro-tumoral effects after thawing. Using a comparative approach, cryopreserved platelets obtained by apheresis were analyzed alongside standard room-temperature stored platelets, currently considered the gold standard for prophylactic transfusion. The protocol involves donor recruitment at the Transfusion Medicine Unit of the AUSL-IRCCS of Reggio Emilia, with platelet concentrates prepared and cryopreserved using 6% dimethyl sulfoxide (DMSO) as well as alternative approaches employing intracellular and extracellular cryoprotectants, either individually or in combination, with lower cytotoxicity reported in other transfusion and cryobiology settings. Platelet samples were evaluated before freezing and after thawing at multiple time points (1, 3, and 6 hours post-reconstitution). Analyses included recovery rate, pH changes, release of bioactive factors, activation markers, hemostatic potential (via thromboelastography), and morphological alterations assessed by flow cytometry, microscopy, and synchrotron-based Fourier transform infrared (FTIR) microspectroscopy. Furthermore, the potential pro-tumoral activity of cryopreserved versus fresh platelets was investigated in vitro using co-culture systems with breast cancer and leukemia cell lines, focusing on proliferation, and platelet-cell interaction tests. The primary objective of this project is to determine the effects of cryogenic storage on platelet function. The secondary objective is to identify the cryopreserved platelet product with the most appropriate safety profile for prophylactic transfusion in onco-hematologic patients. The study is conducted by the BioMetLab at the Transfusion Medicine Unit of AUSL-IRCCS of Reggio Emilia in compliance with the Declaration of Helsinki, following informed consent from all donors.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent

Exclusion Criteria:

* refusal or inability to provide written informed consent

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Platelet donors
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2020-12-31 (Actual); Primary Completion 2021-04-12 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Platelet Recovery Rate After Cryopreservation (Percentage of Initial Count) | through study completion, an average of 4 year
  Platelet recovery will be assessed by calculating the percentage of platelets remaining after cryopreservation compared to pre-freezing values, expressed as recovery rate (%).
Absolute Platelet Count After Cryopreservation (×10⁹/L) | through study completion, an average of 4 year
  Platelet concentration will be determined using an automated hematology analyzer, expressed as absolute platelet count in ×10⁹/L.
Platelet Function Assessed by Thromboelastography - Clot Formation Time | through study completion, an average of 4 year
  Hemostatic function will be analyzed using thromboelastography (TEG). The outcome will include clot formation time (in minutes) as a measure of platelet functional activity.
Platelet Function Assessed by Thromboelastography - Maximum Amplitude | through study completion, an average of 4 years
  Hemostatic function will be analyzed using thromboelastography (TEG). The outcome will include maximum amplitude (in millimeters) as a measure of platelet functional activity.

SECONDARY OUTCOMES:
Release of Pro-Inflammatory Cytokines After Cryopreservation (Concentration in pg/mL) | through study completion, an average of 4 year
  Levels of IL-6 and TNF-α will be quantified in platelet supernatants using ELISA assays, expressed in pg/mL.
Morphological Integrity of Platelets After Cryopreservation (Percentage of Normal Platelets) | through study completion, an average of 4 year
  Morphology will be assessed by light microscopy and flow cytometry, expressed as the percentage of platelets retaining normal morphology.
Hemostatic Potential by Thromboelastography - Clotting Time | through study completion, an average of 4 year
  Hemostatic potential will be evaluated with thromboelastography (TEG). The outcome includes clotting time (in minutes) as a measure of the hemostatic process.
Pro-Tumoral Activity of Cryopreserved Platelets in Co-Culture with Cancer Cell Lines (Percentage Increase in Cell Proliferation) | through study completion, an average of 4 year
  Platelet-tumor interaction will be assessed in vitro using breast cancer and leukemia cell lines. Results will be expressed as the percentage increase in cancer cell proliferation compared to controls.
Hemostatic Potential by Thromboelastography - Maximum Clot Firmness | through study completion, an average of 4 years.
  Hemostatic potential will be evaluated with thromboelastography (TEG). The outcome includes maximum clot firmness (in millimeters) as a measure of clot stability.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda USL IRCCS di Reggio Emilia, Reggio Emilia, Italy

REFERENCES:
- [Background] Ang AL, Gan LSH, Tuy TT, Ang CH, Tan CW, Tan HH, Shu PH, Zhang Q, Cao Y, Moorakonda RB, Pokharkar Y, Lu J. A randomized cross-over study of cryopreserved platelets in prophylactic transfusions of thrombocytopenic patients. Transfusion. 2023 Sep;63(9):1649-1660. doi: 10.1111/trf.17503. Epub 2023 Aug 19. PMID 37596937
- [Background] Christodoulides A, Zeng Z, Alves NJ. In-vitro thromboelastographic characterization of reconstituted whole blood utilizing cryopreserved platelets. Blood Coagul Fibrinolysis. 2021 Dec 1;32(8):556-563. doi: 10.1097/MBC.0000000000001075. PMID 34475333
- [Background] Jimenez-Marco T, Castrillo A, Hierro-Riu F, Vicente V, Rivera J. Frozen and cold-stored platelets: reconsidered platelet products. Platelets. 2022 Jan 2;33(1):27-34. doi: 10.1080/09537104.2021.1967917. Epub 2021 Aug 22. PMID 34423718
- [Background] Reade MC, Marks DC, Howe B, McGuinness S, Parke R, Navarra L, Charlewood R, Johnson L, McQuilten Z; CLIP-II and CLIPNZ-II Investigators.; CLIP-II and CLIPNZ-II Investigators. Cryopreserved platelets compared with liquid-stored platelets for the treatment of surgical bleeding: protocol for two multicentre randomised controlled blinded non-inferiority trials (the CLIP-II and CLIPNZ-II trials). BMJ Open. 2022 Dec 20;12(12):e068933. doi: 10.1136/bmjopen-2022-068933. PMID 36600425
- [Background] Johnson L, Tan S, Wood B, Davis A, Marks DC. Refrigeration and cryopreservation of platelets differentially affect platelet metabolism and function: a comparison with conventional platelet storage conditions. Transfusion. 2016 Jul;56(7):1807-18. doi: 10.1111/trf.13630. Epub 2016 May 9. PMID 27158813
- [Background] Johnson L, Reade MC, Hyland RA, Tan S, Marks DC. In vitro comparison of cryopreserved and liquid platelets: potential clinical implications. Transfusion. 2015 Apr;55(4):838-47. doi: 10.1111/trf.12915. Epub 2014 Nov 5. PMID 25371169
- [Background] Johnson L, Tan S, Jenkins E, Wood B, Marks DC. Characterization of biologic response modifiers in the supernatant of conventional, refrigerated, and cryopreserved platelets. Transfusion. 2018 Apr;58(4):927-937. doi: 10.1111/trf.14475. Epub 2018 Jan 12. PMID 29330877
- [Background] Slichter SJ, Jones M, Ransom J, Gettinger I, Jones MK, Christoffel T, Pellham E, Bailey SL, Corson J, Bolgiano D. Review of in vivo studies of dimethyl sulfoxide cryopreserved platelets. Transfus Med Rev. 2014 Oct;28(4):212-25. doi: 10.1016/j.tmrv.2014.09.001. Epub 2014 Sep 21. PMID 25439164
- [Result] Gavioli G, Razzoli A, Bedolla DE, Di Bartolomeo E, Quartieri E, Iotti B, Berni P, Birarda G, Vaccari L, Schiroli D, Marraccini C, Baricchi R, Merolle L. Cryopreservation affects platelet macromolecular composition over time after thawing and differently impacts on cancer cells behavior in vitro. Platelets. 2023 Dec;34(1):2281943. doi: 10.1080/09537104.2023.2281943. Epub 2023 Nov 27. PMID 38010129